CLINICAL TRIAL: NCT05783921
Title: A Randomized, Open, Multicenter Phase 1/Phase 2 Clinical Trial of TQB2618 Injection Combined With Penpulimab Injection and Chemotherapy Versus Penpulimab Injection Combined With Chemotherapy in First-line Treatment of Relapsed/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Clinical Trial of TQB2618 Injection Combined With Penpulimab Injection and Chemotherapy Versus Penpulimab Injection Combined With Chemotherapy in First-line Treatment of Relapsed/Metastatic Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2618-AK105-Ib-02
Record Dates: First submitted 2023-03-08; First posted 2023-03-24 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Recurrent Squamous Cell Carcinoma of the Head and Neck; Metastatic Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — penpulimab; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2618 injection +Penpulimab injection+Chemotherapy (Paclitaxel+Cisplatin or Carboplatin) (Experimental): TQB2618 injection combined with Penpulimab injection, Paclitaxel, Cisplatin or Carboplatin, 21 days as a treatment cycle. After 4~6 cycles, TQB2618 injection combined with Penpulimab injection, 21 days as a treatment cycle.
  Interventions: Drug: TQB2618 injection, Penpulimab injection, Paclitaxel, Cisplatin or Carboplatin
- Penpulimab injection + Chemotherapy (Paclitaxel+Cisplatin or Carboplatin) (Active Comparator): Penpulimab injection combined with Paclitaxel, Cisplatin or Carboplatin, 21 days as a treatment cycle. After 4~6 cycles, Penpulimab injection, 21 days as a treatment cycle.
  Interventions: Drug: Penpulimab injection, Paclitaxel, Cisplatin or Carboplatin

INTERVENTIONS:
Drug: TQB2618 injection, Penpulimab injection, Paclitaxel, Cisplatin or Carboplatin — TQB2618 injection is an Anti TIM-3 (T-cell immunoglobulin and mucin domain-3) monoclonal antibody.
  Penpulimab injection is a humanized Monoclonal Antibody target Programmed Cell Death Protein 1 (PD-1).
  Paclitaxel is a anti-microtubule drug, which promotes tubulin polymerization, inhibits depolymerization, maintains tubulin stability and inhibits cell mitosis.
  Cisplatin inhibits DNA synthesis by generating in-strand interstrand crosslinking with DNA. Protein and RNA synthesis can also be inhibited.
  Carboplatin is a cyclic nonspecific antitumor agents that cause cross-linking between DNA strands and affect their synthesis to inhibit cancer cells.
  Arms: TQB2618 injection +Penpulimab injection+Chemotherapy (Paclitaxel+Cisplatin or Carboplatin)
Drug: Penpulimab injection, Paclitaxel, Cisplatin or Carboplatin — Penpulimab injection is a humanized Monoclonal Antibody target Programmed Cell Death Protein 1 (PD-1).
  Paclitaxel is a anti-microtubule drug, which promotes tubulin polymerization, inhibits depolymerization, maintains tubulin stability and inhibits cell mitosis.
  Cisplatin inhibits DNA synthesis by generating in-strand interstrand crosslinking with DNA. Protein and RNA synthesis can also be inhibited.
  Carboplatin is a cyclic nonspecific antitumor agents that cause cross-linking between DNA strands and affect their synthesis to inhibit cancer cells.
  Arms: Penpulimab injection + Chemotherapy (Paclitaxel+Cisplatin or Carboplatin)

SUMMARY:
To evaluate the efficacy and safety of TQB2618 injection combined with Penpulimab and chemotherapy in the first-line treatment of relapsed/metastatic head and neck squamous cell carcinoma compared to Penpulimab combined chemotherapy.

Progression-free survival (PFS) and objective response rate (ORR) were the primary efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent form, and had good compliance.
* Between the ages of 18-75 years (calculated based on the date of signing ICF); male or female; Eastern cooperative oncology group (ECOG) score 0-1; estimated survival time ≥ 3 months.
* No indications of local radical therapy for recurrence/metastasis head and neck squamous cell carcinoma.And histologically- or cytologically-confirmed head and neck squamous cell carcinoma ，Primary tumor locations of oropharynx, oral cavity, hypopharynx, or larynx.
* No systemic therapy for recurrent/metastatic lesions, but excluding systemic therapy for locally advanced disease as a part of multimodal therapy (including induction therapy, systemic therapy in the same period of radiotherapy, and adjuvant therapy), and the completion time of treatment was more than 6 months from enrollment (according to the date of informed consent);
* At least one measurable lesion (based on RECIST1.1).
* The main organs function are normally, the following criteria are met:

  1. hemoglobin (Hb) ≥90g/L (no blood transfusion and blood products within 14 days) ；absolute neutrophil count (ANC) ≥1.5×109/L； platelets (PLT) ≥90×109/L.
  2. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN. If accompanied by liver metastases, ALT and AST ≤ 5×ULN; Serum creatinine (CR) ≤ 1.5×ULN or creatinine clearance (CCR) ≥ 60 ml/min.
  3. Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR) ≤ 1.5×ULN (no anticoagulant therapy); Thyroid-stimulating hormone (TSH) ≤ ULN; If abnormalities should be examined, T3 and T4 levels should be examined, and T3 and T4 levels are normal.
  4. Cardiac ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ 50%.
* Female participants of childbearing age should agree to use contraception (e.g., IUDs, pills, or condoms) during the study period and for 6 months after the end of the study; Have a negative serum pregnancy test within 7 days prior to study enrollment and must be a non-lactating subject; Male participants should agree that contraception must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Comorbidity and medical history:

  1. Have had or currently have other malignant tumors within 3 years. The following two conditions can be enrolled: other malignancies treated with a single surgery to achieve 5-year disease-free survival (DFS); cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumors), Tis (carcinoma in situ) and T1 (tumor-invasive basement membrane)];
  2. adverse effects due to any prior treatment have not been restored to CTCAE 5.0 ≤ level 1 (except for toxicity where the investigator determines that there is no safety risk);
  3. Major surgical treatment, incision biopsy, or significant traumatic injury were received within 28 days prior to study treatment
  4. Long-term unhealed wounds or fractures
  5. Arteriovenous thrombotic events within 6 months, such as cerebrovascular accidents;
  6. Those who have a history of psychotropic substance abuse and cannot quit or have a mental disorder;
  7. Subjects with any severe and/or uncontrolled medical conditions, including:

     1. Unsatisfactory blood pressure control (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥100 mmHg);
     2. Have grade ≥2 myocardial ischemia or myocardial infarction, arrhythmias (including QTc ≥ 450 ms (male) in men and QTc ≥ 470 ms (female)) and grade ≥ congestive heart failure grade 2 (New York Heart Association (NYHA) grade);
     3. Active or uncontrolled severe infection (≥ CTC AE grade 2 infection) or unexplained fever > 38.5°C;
     4. Liver cirrhosis, active hepatitis Note: Active hepatitis (hepatitis B reference: HBsAg positive and HBV (hepatitis B virus) DNA detection value of more than 1000 copies /mL; Hepatitis C reference: HCV (hepatitis C virus) antibody positive, and HCV virus titer test value above the upper limit of normal);
     5. Known to have syphilis;
     6. Renal failure requires hemodialysis or peritoneal dialysis
     7. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
     8. Poor diabetes control [fasting blood glucose (FBG) > 10mmol/L]
     9. Urine routine indicated urine protein ≥++, and confirmed 24 hours urine protein quantity > 1.0 g
     10. People who have epilepsy and need treatment
* Tumor related symptoms and treatment

  1. Study history of surgery, chemotherapy, radiotherapy, or other anticancer therapy within 4 weeks prior to the start of treatment (washout period from the end of the last treatment)；
  2. progress during or within 6 months of completion of systemic therapy (including induction therapy, concurrent radiotherapy, adjuvant therapy) for locally advanced disease;
  3. Secondary radiotherapy was performed for local recurrent lesions;
  4. Received Chinese patent drugs with anti-tumor indications specified in the Chinese National Medical Product Administration approved drug instructions within 1 week before the study treatment;
  5. Have received relevant immunotherapy drugs in the past;
  6. where imaging (CT or MRI) shows that the tumor has invaded important blood vessels, or the investigator determines that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during the follow-up study period;
  7. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (investigator's judgment)
  8. Subjects with known central nervous system metastatic and/or cancerous meningitis;
* Research and treatment related:

  1. Study history of live attenuated vaccine vaccination within 28 days before the start of treatment or planned live attenuated vaccine vaccination during the study period;
  2. Patients with a definite tendency to bleed or clinically significant bleeding symptoms, including but not limited to gastrointestinal bleeding, nasal bleeding, and hemorrhagic disease or coagulopathy within 28 days prior to initial medication;
  3. People who have experienced severe hypersensitivity after the use of monoclonal antibodies, or are allergic to known components of the drug under study;
  4. Study of active autoimmune diseases requiring systemic treatment that occurred within 2 years prior to initiation of treatment;
  5. Have been diagnosed with immunodeficiency or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose > 10mg/ day prednisone or other efficacy hormone) and continue to use within 2 weeks before the study therapy begins;
* Participated in clinical trials of other antitumor drugs within 4 weeks before the first medication;
* Subjects who, in the judgment of the investigator, have concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are not suitable for inclusion for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Baseline to up to two years.
  The time period from the first administration of the drug to disease progression or death event (whichever occurs first).
Objective response rate (ORR) | Baseline to up to two years.
  According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and iRECIST, the proportion of subjects whose tumors are evaluated as complete response(CR) and partial response(PR) by subcenter imaging evaluation. It is recorded from the first administration of the drug to disease progression or initiation of a new anticancer treatment.

SECONDARY OUTCOMES:
PFS rate at 9 months | Baseline to 9 months
  Proportion of survived participants without progression at 9th months.
Overall survival (OS) | Baseline to up to two years.
  Time from the randomization to death from all causes.
Disease Control Rate (DCR) | Baseline to up to two years.
  The percentage of participants with complete response (CR), partial response (PR), or stable disease (SD) for 6 weeks or more as determined by investigators according to RECIST 1.1.
Clinical benefit rate (CBR) | Baseline to up to two years.
  The percentage of participants with complete response (CR), partial response (PR), or stable disease (SD) for 6 months or more as determined by investigators according to RECIST 1.1.
Duration of Remission (DOR) | Baseline to up to two years.
  The period from firstly-recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurs first).
Incidence of adverse events (AEs) | Baseline to up to two years.
  All adverse medical events that occur after the subject receives the investigational drug may be manifested as symptoms, signs, disease, or laboratory abnormalities, but are not necessarily causally related to the investigational drug, evaluated according to the National Cancer Institute standard for common toxic criteria [NCI-CTC v5.0].
Severity of adverse events (AEs) | Baseline to up to two years.
  All adverse medical events that occur after the subject receives the investigational drug may be manifested as symptoms, signs, disease, or laboratory abnormalities, but are not necessarily causally related to the investigational drug, evaluated according to the National Cancer Institute standard for common toxic reactions [NCI-CTC v5.0].
Serious adverse events (SAEs) | Baseline to up to two years.
  It refers to adverse medical events such as death, life-threatening, permanent or serious disability or loss of function, hospitalization or prolonged hospitalization, and congenital abnormalities or birth defects after the subject receives the experimental drug.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Gansu Prouincial Cancer Hospital, Lanzhou, Gansu
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - AnYang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhumadian Centre Hospital, Zhumadian, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Liaoning Cancer hospital, Shenyang, Liaoning
  - The Second Hospital Of Dalian Medical University, Shenyang, Liaoning